CLINICAL TRIAL: NCT02466152
Title: A Pharmacokinetic Study for Systemic Exposure of Twice Daily Topically Applied GSK2894512 Cream in Subjects With Atopic Dermatitis
Brief Title: Pharmacokinetic Study of Topical GSK2894512 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201851
Record Dates: First submitted 2015-05-21; First posted 2015-06-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dermatitis, Atopic
Keywords: PK; GSK2894512; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2894512 2.0% Cohort (Experimental): Subjects will apply a thin layer of GSK2894512 2.0% topical cream twice daily (morning and evening) for 20 days and only in morning on day 21, to all affected skin areas (15-35% BSA) identified at baseline, excluding the scalp and around the eyes
  Interventions: Drug: GSK2894512 Topical Cream
- GSK2894512 1.0% Cohort (Experimental): Subjects will apply a thin layer of GSK2894512 1.0% topical cream twice daily (morning and evening) for 20 days and only in morning on day 21, to all affected skin areas (15-35% BSA) identified at baseline, excluding the scalp and around the eyes
  Interventions: Drug: GSK2894512 Topical Cream

INTERVENTIONS:
Drug: GSK2894512 Topical Cream — GSK2894512 will be supplied as white to off-white topical cream in doses of 2.0% (20 milligrams/gram [mg/g]) and 1.0% (10 mg/g)

SUMMARY:
This study will assess the systemic exposure and pharmacokinetic parameters of GSK2894512 following twice daily topical administration of 1% and 2% cream in adult subjects with AD, and will provide information about the systemic safety as well as local safety and tolerability following twice daily application to up to 35% body surface area (BSA) of affected skin of subjects with AD. It will be an open-label, sequential study consisting of 2 cohorts. A cohort of 6 subjects (Cohort 1) will apply GSK2894512 (cream, 2%) to affected skin on an area ranging from 15 to 35% of the total BSA for 20 days plus a final dose on Day 21. Cohort 2 will consist of 6 subjects that will apply 1% cream. Cohort 2 will follow the same procedures as Cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Confirmed clinical diagnosis of AD according to established criteria by Hanifin at the screening visit.
* History of AD of at least 6 months.
* Atopic dermatitis on 15-35%, of the BSA, (scalp and area around the eyes not included as treatment area) at baseline. Note: 1% BSA is approximately equal to the surface of one hand with fingers together (a handprint)
* An IGA of AD score of >=3 at baseline.
* Male: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least five half-lives of study medication after the last dose of study medication:

  1. Vasectomy with documentation of azoospermia.
  2. Male condom plus partner use of one of the contraceptive options: Contraceptive sub-dermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone, Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* A woman is eligible to participate if she is of non-reproductive potential, defined as:

  1. Postmenopausal (including all women over 60 years of age).
  2. Females with one of the following procedures documented and no plans to utilize assisted reproductive techniques (e.g., in vitro fertilization or donor embryo transfer): Bilateral tubal ligation or salpingectomy; Hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Bilateral oophorectomy (surgical menopause) Note: A practical definition accepts menopause after 1 year without menses with an appropriate clinical profile (e.g., age appropriate, >45 years, in the absence of hormone replacement therapy [HRT] or medical suppression of the menstrual cycle). In questionable cases for women <60 years of age, a blood sample with simultaneous follicle stimulating hormone and estradiol falling into the central laboratory's postmenopausal reference range is confirmatory. Women <60 years of age who are on HRT, wish to continue, and whose menopausal status is in doubt are required to use a highly-effective method to avoid pregnancy. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of postmenopausal status, HRT may be resumed during the study without use of a highly-effective method to avoid pregnancy
* Capable of giving signed informed consent as described in Protocol which includes compliance with the requirements and restrictions listed in the consent form and in protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTc > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block.

NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).

* Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to dosing (Day 1).
* Chronic or acute infection requiring treatment with systemic treatments (antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals) within 4 weeks before dosing, or superficial skin infections within 1 week before the screening visit.
* Concurrent conditions and history of other diseases: Immunocompromized (e.g., lymphoma, Acquired Immuno Deficiency Syndrome, Wiskott-Aldrich Syndrome) or have a history of malignant disease within 5 years before the baseline visit; Presence at screening or baseline of an active acute bacterial, fungal or viral skin infection (e.g., herpes simplex, herpes zoster, chicken pox); Any other concomitant skin disorder (e.g., generalized erythroderma such as Netherton's Syndrome, or psoriasis), significant hyperpigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise subject safety; Clinical signs of infection (viral, fungal or bacterial) on the treatment areas; Other types of eczema.
* Used any prohibited medication listed in Protocol within the indicated washout period
* Prolonged exposure to natural or artificial sources of ultraviolet (UV) radiation that results in sunburn within 2 weeks prior to the first dose
* And/or intention to have UV exposure during the study, which is thought by the investigator to be likely to modify the subject's AD.
* Planning to use a sauna during the duration of the study or intending to swim
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive drug/alcohol screen at screening.
* A positive test for Human immunodeficiency virus (HIV) antibody at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* A history or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* Use of anti-coagulant medication (e.g. heparin, Low Molecular Weight -heparin, warfarin, anti-platelets [Nonsteroidal anti-inflammatory drugs and low dose aspirin 81 milligrams will not be considered anti platelets]) or a contraindication to skin biopsies, a history of hypertrophic scarring or keloid formation in scars or suture sites, or a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
* Use of nicotine-containing products (including nicotine patches).
* Women who are pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2015-10-27 (Actual); Study Completion 2015-10-27 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters | On Day 1 at pre-dose, 1 hour (h), 2h, 4h, 8h, 10h, 12h, 14h, 16h; On Days 2, 3, 4, 7 and 14 at Pre-dose; On Day 21 at pre-dose, 1h, 2h, 4h, 8h, 10h, 12h; On Day 22 at 0h
  PK parameters include plasma concentrations of GSK2894512, maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve (AUC) to last measurable concentration [AUC(0-t)], AUC through 24 hours [AUC(0-24)] and AUC per dosing interval [AUC(0-tau)], apparent terminal phase half-life following the last dose (t1/2); steady-state trough concentrations (Ctau), accumulation ratio (Ro), as data allows.
Number of subjects with adverse events (AEs) | Up to Day 22
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product temporally associated with the use of a medicinal product
Safety as assessed by Vital signs | Up to Day 22
  Vital signs will include height (only at baseline) and weight (only at baseline and Day 22), temperature, systolic and diastolic blood pressure and pulse rate
Safety as assessed by electrocardiogram (ECG) parameters | Up to Day 22
  Triplicate 12-lead ECGs will be obtained at each time-point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals.
Safety as assessed by abbreviated physical examination parameters | Baseline and Day 22
  Physical examination will include assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
Safety as assessed by clinical laboratory assessments | Baseline, Day 7, 14 and Day 22
  Clinical laboratory assessments will include hematology, clinical chemistry, urinalysis parameters
Local tolerability as assessed by degree of local irritation | Baseline , Days 1, 2, 3, 4, 7, 14, 21 and 22
  The application sites will be assessed for presence and overall degree of irritation

SECONDARY OUTCOMES:
Change from baseline in Eczema Area and Severity Index (EASI) | Baseline (Day -1) and Days 3, 7, 14 and 21
  The EASI scoring system is a standard clinical tool for assessing the severity of AD that takes into account the overall severity of erythema, infiltration/papulation, excoriation, and lichenification, as well as the extent of BSA affected with AD.
Proportion of subjects with >=50% improvement in EASI | Baseline (Day -1) and Days 3, 7, 14 and 21
Proportion of subjects who achieve an Investigator's Global Assessment (IGA) of 0 or 1 and have at least a 2-point improvement over baseline | Baseline (Day -1) and Days 3, 7, 14 and 21
  IGA is a clinical tool for assessing the current state/severity of the subject's AD.
Change from baseline in subject's pruritus (numeric rating scale [NRS]) | Baseline and up to Day 22
  Subject-reported itch (pruritus) severity will be analyzed by the daily sign and symptom severity diary NRS.
Change from baseline in % BSA affected | Baseline (Day -1) and Days 3, 7, 14 and 21
  Percentage of body surface area (BSA) affected will be assessed at the specified time points.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bissonnette R, Vasist LS, Bullman JN, Collingwood T, Chen G, Maeda-Chubachi T. Systemic Pharmacokinetics, Safety, and Preliminary Efficacy of Topical AhR Agonist Tapinarof: Results of a Phase 1 Study. Clin Pharmacol Drug Dev. 2018 Jun;7(5):524-531. doi: 10.1002/cpdd.439. Epub 2018 Feb 1. PMID 29389078
- See also: Results for study 201851 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201851?search=study&b'study_ids=201851'#rs